CLINICAL TRIAL: NCT05691348
Title: Same Day Ambulatory Appendectomy (SAMBA)
Acronym: SAMBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-API-01
Record Dates: First submitted 2023-01-09; First posted 2023-01-20 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulatory pathway (Experimental)
  Interventions: Procedure: Ambulatory appendectomy
- Conventional hospitalisation (Active Comparator)
  Interventions: Procedure: Conventional appendectomy

INTERVENTIONS:
Procedure: Ambulatory appendectomy — Appendectomy will be performed in outpatient surgery unit. Patient will be discharge from the hospital the same day as surgery
  Arms: Ambulatory pathway
Procedure: Conventional appendectomy — Appendectomy will be performed in digestive surgery department. Patient will be discharge from the hospital the day after surgery: he will spend a night under observation
  Arms: Conventional hospitalisation

SUMMARY:
The potential benefit of outpatient care for this common digestive emergency is considerable, both for the patients themselves and for the public health system:

1. Optimization of the care pathway, reducing the length of stay in hospital (a major issue in the context of the COVID-19 (coronavirus disease) pandemic) liberating patient beds and staff, and reducing the risk of nosocomial exposure.
2. Improved patient satisfaction compared to waiting for hours in the emergency department due to lack of hospital beds.
3. Non-inferiority of care in an outpatient unit in terms of quality and safety in day hospitalization.
4. Significant decrease in the overall cost of this pathology as a result of a reduction in the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15-74 years
* BMI ≤ 30 kg/m2
* Uncomplicated acute appendicitis confirmed by imaging (ultrasound and/or CT and/or MRI)

  * Temperature ≤ 38,1°C and > 35,5°C
  * Appendix diameter > 6mm and ≤ 15mm
  * Without effusion or with only localized peri-appendicular effusion
  * Infiltration of peri-appendicular fat without abscess or plastron
  * No sign of perforation
  * Leukocytes ≤ 15,000G/L AND
  * CRP (C reactive protein) ≤ 50mg/L
* If pain, calmed by level 2 analgesic at maximum
* Ambulatory criteria

  * Availability of monitoring by a relative during the 12 hours after discharge from the hospital
  * Residence located less than 20 minutes by car from a health center (hospital or clinic)
  * Access to a telephone mobile or fixed in case of problems
* Signature of the written informed consent form by the patient
* If the patient is a minor, signature of the written informed consent form by both parents or their legal representative
* Affiliation to a French health insurance scheme or equivalent

Exclusion Criteria:

* Criteria that exclude ambulatory care such as an ASA score (Physical status score) > 2, severe or uncontrolled comorbidities, severe pulmonary disease including obstructive sleep apnea, anticoagulation or antiplatelet drug or contraindication to ambulatory surgery such as intubation difficulties
* Presence of active cancer, a malignant hemopathy, drug addiction, coagulopathy, immunosuppressive treatment
* Non-acute or interval appendectomy, i.e. after antibiotic treatment of a complicated appendicitis of the plastron or drainage of an appendicular abscess;
* History of pelvic surgery
* Vulnerable people: pregnant or breast-feeding women (patients will undergo a pregnancy test: plasmatic β-hCG (human chorionic gonadotropin) or urinary test), adult under guardianship or deprived of freedom. Pregnant women are considered to have a full stomach, with risk of inhalation at anesthetic induction and represent a contraindication to ambulatory surgery. In addition, the need to perform abdominal surgery on a pregnant woman requires obstetric monitoring that is difficult to reconcile with management in an outpatient surgery unit (need for obstetric ultrasound or monitoring).
* Suspicion of a tumor of the appendix : Mucocele and pseudomyxoma, Carcinoid tumor, Adenocarcinoma of the appendix, Another type of tumor

Ages: 15 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that outpatient care, compared with conventional care, in selected patients with acute uncomplicated appendicitis operated by laparoscopy, is non-inferior in terms of overall morbi-mortality on the 30th postoperative day. | 30 days post surgery
  Morbi-mortality will be assessed by classifying post-operative complications according to Clavien-Dindo classification. It will be compared between both groups ("ambulatory pathway" versus "conventional hospitalization" CONV) on the 30th postoperative day.
  The Clavien-Dindo classification was originally published in 2004 in the Annals of Surgery for elective general surgery. Later, it has been objectively validated for all surgical specialties. This classification ranks complications from 0 (no complication) to 5 (death). Complications that potentially lead to long-lasting disability after discharge (e.g.: paralysis of a vocal cord after thyroid surgery) are highlighted in the present classification by a suffix ("d" for disability). This suffix indicates that a long-term follow-up is required to comprehensively evaluate the outcome and related long-term quality of life.

SECONDARY OUTCOMES:
To compare between both groups, at post-operative day 30, the delay from diagnosis to appendectomy | 30 days post surgery
  The delay from diagnosis to appendectomy is defined as the time between the performance of the CT scan (or ultrasound or MRI) for diagnosis and the skin incision in the operating room. This time is expressed in minutes.
To compare between both groups, at post-operative day 30, the real cumulated length of hospitalization | 30 days post surgery
  The real cumulated length of hospitalization is the cumulative length of the entire hospital stay(s) in hours until the 30th postoperative day (rehospitalizations included). The length of stay in a non-hospital health structure, such as a convalescent center, will not be included.
To compare between both groups, at post-operative day 30, the rehospitalization rate | 30 days post surgery
  All re-hospitalization(s) after initial discharge will be counted until 30 days post surgery, whatever the cause or type of hospitalization.
To compare between both groups, the mild morbidity (Clavien-Dindo I-II) during 30 days post surgery | up to the 30th day post surgery
  Post-operative mild morbidity will be assessed with the Clavien-Dindo classification (grade I, II) up to the 30th day post surgery. Clavien-Dindo classification was originally published in 2004 in the Annals of Surgery for elective general surgery. Later, it has been objectively validated for all surgical specialties. This classification ranks complications from 0 (no complication) to 5 (death).
To compare between both groups, the severe morbidity (Clavien-Dindo III, IV, V) during 30 days post surgery | up to the 30th day post surgery
  Post-operative mild morbidity will be assessed with the severe morbidity (Clavien-Dindo III, IV, V) up to the 30th day post surgery. Clavien-Dindo classification was originally published in 2004 in the Annals of Surgery for elective general surgery. Later, it has been objectively validated for all surgical specialties. This classification ranks complications from 0 (no complication) to 5 (death).
To compare between both groups, the rate of interventional radiology re-intervention (radio-guided drainage) | up to the 30th day post surgery
  All the Clavien-Dindo interventional radiology re-interventions (radio-guided drainage) performed in relation with the appendicitis and any potential complications will be recorded up to the 30th day post surgery.
To compare between both groups, the rate of laparoscopic re-intervention | up to the 30th day post surgery
  All laparoscopic re-interventions performed in relation with the appendectomy and the potential complications will be recorded up to the 30th day post surgery.
To compare between both groups, at post-operative day 30, the rate of re-intervention by laparotomy | up to the 30th day post surgery
  All the laparotomic re-interventions performed in relation with the appendectomy and the potential complications will be recorded up to the 30th day post surgery.
To compare between both groups, patient satisfaction 7 and 30 days post surgery | 7 and 30 days post surgery
  Patient satisfaction will be assessed using a numerical scale from 0 to 10, using the Link4Life app. Zero '0', placed on the left, means that the patient is not satisfied at all with her/his postoperative course; '10', placed on the right, means that the patient is extremely satisfied with her/his postoperative course. If the patient does not have access or does not wish to access Link4Life, a clinical research assistant from the investigating center will collect the patient's satisfaction through a phone call. The questions that will be asked are: "How satisfied are you with your care?"; "are you in pain and if so, how severe is it?"; "Were you worried about same-day discharge (for patients in the outpatient group)?
To compare between both groups, patient quality of life 7 and 30 days post surgery | at inclusion and at 7 and 30 days post surgery
  Quality of life will be evaluated using the EuroQol five-dimension questionnaire (EQ-5D-5L), at inclusion, and at 7 and 30 days post surgery.The EQ-5D-5L comprises a descriptive system and a visual analogue scale (VAS). The descriptive system is composed of five health dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with 5 levels of health (no problems, slight problems, moderate problems, severe problems and extreme problems). For each of the 5 dimensions, the participant's answer is converted to a number between 1 and 5, expressing the health state reported. The responses are combined to produce a five-digit number describing the participant's health status which is converted to a utility value from the country specific value set. The French EQ-5D-5L value set has utility between -0.530 (health condition worse than death) and 1 (best possible health). The VAS records the self-rated health status on a graduated scale from 0 to 100.
To evaluate the rate of conversion from outpatient to conventional care | up to the 30th day post surgery
  A conversion will be defined as a patient randomized to the outpatient care group who is finally treated following the conventional care procedure, whatever the reason
To estimate the cost of outpatient appendectomy management | up to the 30th day post surgery
  The cost will be estimated by the hospital cost (intervention and outpatient stay).
To study the economic impact (utility) of outpatient appendectomy management compared to conventional hospitalization | up to the 30th day post surgery
  The economic impact will be studied with a cost-utility analysis which will estimate the incremental cost-effectiveness ratio (ICER) in cost per QALY (quality adjusted life years) gained.
To study the economic impact (effectiveness) of outpatient appendectomy management compared to conventional hospitalization | up to the 30th day post surgery
  The economic impact will be studied with a cost-effectiveness analysis which will estimate the ICER in cost per patient without rehospitalization.
To study the generalization of outpatient appendectomy management in all French hospitals at the budgetary level | up to the 30th day post surgery
  The generalization of outpatient appendectomy management will be studied with a budget impact model which will estimate the consequences in terms of costs
To study the generalization of outpatient appendectomy management in all French hospitals at a strategic level | up to the 30th day post surgery
  The generalization of outpatient appendectomy management will be studied with QALYs (quality adjusted life years) of the adoption of the outpatient strategy in all French hospitals

CONTACTS AND LOCATIONS:
Locations (33):
- France (31):
  - Hôpitaux Pédiatriques de Nice CHU - Lenval, Nice, Alpes Maritimes
  - CHU de Nice, Nice, Alpes-Maritimes
  - CHU de Bordeaux, Bordeaux, Aquitaine
  - CH de Troyes, Troyes, Aube
  - CHU Grenoble Alpes, La Tronche, Auvergne-Rhône-Alpes
  - Hôpital Edouard HERRIOT, Lyon, Auvergne-Rhône-Alpes
  - CHU de Saint-Etienne - Hôpital Nord, Saint-Priest-en-Jarez, Auvergne-Rhône-Alpes
  - CH de Voiron, Voiron, Auvergne-Rhône-Alpes
  - APHM Hôpital Nord, Marseille, Bouches-du-Rhône
  - CHU Minjo, Besançon, Bourgogne-Franche-Comté
  - CHU de Rennes, Rennes, Brittany Region
  - Hôpital Robert Debré - CHU de Reims, Reims, Grand Est
  - Hôpital Beaujon (APHP), Clichy, Hauts De Seine
  - CHU Amiens-Picardie, Amiens, Hauts-de-France
  - Clinique de Saint-Omer, Blendecques, Hauts-de-France
  - HIA Percy, Clamart, Hauts-de-Seine
  - CHU de Tours, Tours, Indre Et Loire
  - CHU de Reims, Reims, Marne
  - CH de Dax, Dax, Nouvelle-Aquitaine
  - CH de Mont de Marsan, Mont-de-Marsan, Nouvelle-Aquitaine
  - CHU d'Angers, Angers, Pays de la Loire Region
  - Hôpital d'Instruction des armées Laveran, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital d'Instruction des armées Sainte Anne - BCRM Toulon, Toulon, Provence-Alpes-Côte d'Azur Region
  - Clinique du Val d'Ouest, Écully, Rhones-Alpes
  - Hôpital Cochin APHP, Paris
  - Hôpital Avicenne, Bobigny, Île-de-France Region
  - Hôpital Louis-Mourier, Colombes, Île-de-France Region
  - APHP Pitié Salpetrière, Paris, Île-de-France Region
  - APHP Lariboisière, Paris, Île-de-France Region
  - Hia Begin, Saint-Mandé, Île-de-France Region
  - Clinique de l'Estrée, Stains, Île-de-France Region
- Reunion (2):
  - CHU de La Réunion, Saint-Denis, La Réunion
  - CHU de La Réunion, Saint-Pierre, La Réunion

REFERENCES:
- [Derived] Arvieux C, Tidadini F, Barbois S, Fontas E, Carles M, Gridel V, Orban JC, Quesada JL, Foote A, Cruzel C, Anthony S, Bulsei J, Hivelin C, Massalou D. SAME day amBulatory c (SAMBA): a multicenter, prospective, randomized clinical trial protocol. Trials. 2024 Sep 9;25(1):601. doi: 10.1186/s13063-024-08336-x. PMID 39252106